CLINICAL TRIAL: NCT06739395
Title: A Pan-Cancer Basket, Real World, Open-label, Multicenter Study on Molecular Matching Therapy Guided by Molecular Tumor Boards (MTB) for Pan Solid Tumor Patients With Standard Treatment Exhaustion
Brief Title: Precision Medicine Trial Based on Molecular Matching Therapy for Patients With Standard Treatment Exhaustion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MyCustom-02
Record Dates: First submitted 2024-12-08; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor; Precision Medicine
MeSH Terms: interventions — olaparib; Temozolomide; anlotinib; trametinib; dabrafenib; Alpelisib; lenvatinib; pazopanib; palbociclib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Monotherapy (Other): In the OncoKB(Precision Oncology Knowledge Base) database, the gene alteration has a variant of clinical evidence in this tumor or other tumor types and is considered to be an interventional variant. Cohort-1may include different observation subgroups（dMMR/MSI-H,TMB-H,NTRK fusion,RET-fusion,BRAF(p.V600E),KRAS(p.G12C),HER2(IHC,3+)）. For example, substudy-1: monotherapy/combination therapy for patients with A1-relative. Substudy-x: monotherapy/combination therapy for patients with Ax-relative.
  Interventions: Drug: Target Gene
- Combination therapy-cohort1 (Experimental): The characteristics of enrolled patients are the presence of two or more interventional or potential actionable targets(only TP53 alteration,MAP2K1 alteration,PMA pathway alteration,11q13 amplification,MET alteration).
  Interventions: Drug: Olaparib tablet; Drug: Temozolomide capsule; Drug: Anlotinib; Drug: Trametinib tablet; Drug: Dabrafenib; Drug: Vebreltinib Enteric Capsules; Drug: Alpelisib Pill; Drug: Sacituzumab Govitecan-Hziy 180 MG; Drug: Lenvatinib Capsules; Drug: Pazopanib Pill; Drug: Palbociclib Pill; Drug: Chidamide; Drug: PD-1/PD-L1/PD-1&CTLA4 inhibitor; Drug: Target Gene
- Combination therapy-cohort2 (Experimental): The characteristics of enrolled patients are primary or secondary drug resistance during treatment.
  Interventions: Drug: Olaparib tablet; Drug: Temozolomide capsule; Drug: Anlotinib; Drug: Trametinib tablet; Drug: Dabrafenib; Drug: Vebreltinib Enteric Capsules; Drug: Alpelisib Pill; Drug: Sacituzumab Govitecan-Hziy 180 MG; Drug: Lenvatinib Capsules; Drug: Pazopanib Pill; Drug: Palbociclib Pill; Drug: Chidamide; Drug: PD-1/PD-L1/PD-1&CTLA4 inhibitor; Drug: Target Gene
- Olaparib+Anlotinib/Temozolomide (Experimental): The gene TP53 alteration that MTB combines with clinical practice and literature reports that can match targeted therapy is considered to be potential actionable targets.
  Interventions: Drug: Olaparib tablet; Drug: Temozolomide capsule; Drug: Anlotinib
- Trametinib±Vebreltinib (Experimental): The gene MAP2K1 alteration that MTB combines with clinical practice and literature reports that can match targeted therapy is considered to be potential actionable targets.
  Interventions: Drug: Trametinib tablet; Drug: Dabrafenib
- Alpelisib (Experimental): The PMA(PI3K/mTOR/AKT ) pathway active alteration that MTB combines with clinical practice and literature reports that can match targeted therapy is considered to be potential actionable targets.This subgroup is not included in breast cancer patients.
  Interventions: Drug: Alpelisib Pill
- Palbociclib+Pazopanib (Experimental): The gene alteration(Chromosome 11q13 amplification (CCND1, FGF3, FGF4, and FGF19)) that MTB combines with clinical practice and literature reports that can match targeted therapy is considered to be potential actionable targets.
  Interventions: Drug: Pazopanib Pill; Drug: Palbociclib Pill
- Vebreltinib (Experimental): MET inhibitors have recently demonstrated clinical activity in patients with MET exon 14 (METex14)-skipping/MET-amplification.
  Interventions: Drug: Vebreltinib Enteric Capsules
- Combination therapy group based on PD-1/L1 immune checkpoint inhibitors (Experimental): MTB combined with clinical practice and literature reports can not match the gene alteration of targeted therapy, which is considered as an irreversible gene alteration.This subgroup may use functional models (including but not limited to PDX(Patient-Derived Tumor Xenograft Model), organoids, etc.) for intervention therapy.
  Interventions: Drug: Lenvatinib Capsules; Drug: Chidamide; Drug: PD-1/PD-L1/PD-1&CTLA4 inhibitor; Drug: Target Gene

INTERVENTIONS:
Drug: Olaparib tablet — Usage and dosage: The recommended dosage is 200mg, twice a day, equivalent to a total daily dose of 400mg.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided(from the I-PREDICT study).
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Olaparib+Anlotinib/Temozolomide
Drug: Temozolomide capsule — Administration method and dosage: 75mg/m2, orally administered for 7 consecutive days, with a treatment cycle of every 21 days.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Olaparib+Anlotinib/Temozolomide
Drug: Anlotinib — Usage, dosage, and administration method: Take orally once a day before breakfast. Take the medication continuously for 2 weeks and stop taking it for 1 week, that is, 3 weeks (21 days) is one course of treatment. Until disease progression or intolerable toxic side effects occur.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Olaparib+Anlotinib/Temozolomide
Drug: Trametinib tablet — Usage, dosage, and administration method: The recommended dose is 2 mg, taken orally once a day with an interval of approximately 24 hours. The dose should be taken at least 1 hour before meals or 2 hours after meals. Do not take any missed doses of trametinib within 12 hours of taking the next dose.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Trametinib±Vebreltinib
Drug: Dabrafenib — Usage and dosage: Take 150mg orally twice a day, with an interval of about 12 hours.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided. When this product is used in combination with trametinib, it should be taken once a day at the same time, along with this product administered in the morning or evening.The dosage for combined use will be adaptively adjusted by the researcher.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Trametinib±Vebreltinib
Drug: Vebreltinib Enteric Capsules — Usage and dosage: The recommended starting dose is 200 mg/time, taken orally twice a day (once in the morning and once in the evening), until disease progression or intolerable toxicity occurs.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Vebreltinib
Drug: Alpelisib Pill — Usage and dosage: The recommended dosage is 300mg (two 150mg film tablets), taken once a day with food; Continue treatment until the disease worsens or unacceptable toxicity occurs.Administration method: Patients should take aspirin at approximately the same time every day and swallow the entire aspirin tablet (the tablet should not be chewed, crushed, or separated before swallowing).The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Alpelisib; Combination therapy-cohort1; Combination therapy-cohort2
Drug: Sacituzumab Govitecan-Hziy 180 MG — Usage and dosage: The recommended dosage is 10 mg/kg, administered intravenously every 21 days as a treatment cycle on the 1st and 8th days, and continued until disease progression or unacceptable toxicity occurs. The dosage of this product should not exceed 10 mg/kg.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2
Drug: Lenvatinib Capsules — Usage and dosage: For patients weighing less than 60kg, the recommended daily dose of lenvatinib is 8mg once a day; For patients weighing ≥ 60kg, the recommended daily dose of lenvatinib is 12mg once daily. Lunvatinib should be taken at a fixed time every day, on an empty stomach or with food.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy group based on PD-1/L1 immune checkpoint inhibitors; Combination therapy-cohort1; Combination therapy-cohort2
Drug: Pazopanib Pill — Usage and dosage: In the safety introduction section, the initial dose of pazopanib is 400mg, and in the dose escalation queue, the dose of pazopanib is 600mg.The dosage for combined use will be adaptively adjusted by the researcher.
  Administration method: Oral treatment once a day, with a cycle of 28 days.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Palbociclib+Pazopanib
Drug: Palbociclib Pill — Usage, dosage, and administration method: 100mg, orally administered once daily for 21 consecutive days, followed by a 7-day discontinuation; Every 28 days is a treatment cycle.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy-cohort1; Combination therapy-cohort2; Palbociclib+Pazopanib
Drug: Chidamide — Usage and dosage: It is recommended to take 30mg (6 tablets) each time, twice a week, with an interval of no less than 3 days between each dose (such as Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.). It should be taken 30 minutes after breakfast.The dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy group based on PD-1/L1 immune checkpoint inhibitors; Combination therapy-cohort1; Combination therapy-cohort2
Drug: PD-1/PD-L1/PD-1&CTLA4 inhibitor — Refer to the respective instructions for use, and the dosage for combined use will be adaptively adjusted by the researcher.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy group based on PD-1/L1 immune checkpoint inhibitors; Combination therapy-cohort1; Combination therapy-cohort2
Drug: Target Gene — Granting CFDA or FDA approved drugs(off-label approved drugs) based on specific molecular characteristics.Essentially, for de novo combinations, we started patients at about 50% of the usual dose of each drug for two-drug combinations, and at about one-third of the dose of each drug for three-drug combinations. Patients then received escalating doses of drugs to tolerance, while being monitored closely by their treating physicians. Combinations of drugs with overlapping toxicities were avoided.
  Arms: Combination therapy group based on PD-1/L1 immune checkpoint inhibitors; Combination therapy-cohort1; Combination therapy-cohort2; Monotherapy

SUMMARY:
The main purpose of this study is to explore the feasibility of selecting treatment plans based on genomic variations guided by MTB in patients with advanced refractory solid tumors.

DETAILED DESCRIPTION:
Using comprehensive genome sequencing to analyze recurrent and metastatic solid tumors that have failed previous conventional treatments, and matching possible targeted therapy drugs to screen for potential effective treatment drugs until tumor disease progression, and then continuing to monitor tumor resistance mutation signals and provide matching therapy, can help improve the clinical outcomes of patients with advanced refractory tumors, and is also an important direction for personalized and precise treatment of tumors in the future. Therefore, the investigators designed this study to explore the feasibility, effectiveness, and safety of targeted therapy based on tumor molecular feature matching for advanced solid tumor patients who have failed previous treatments. All patients who receive treatment with a drug available in the protocol will be followed for standard efficacy outcomes including clinical efficacy ,clinical safety and exploratory endpoints such as biomarkers for drug response, change in the tumor microenvironment. The core concepts of the clinical research interventional initiated include: target priority principle, combination therapy principle, individualized dose adjustment method for combination therapy, and Bayesian adaptive trial design. For some clinical studies, to meet the primary objective, at least 35% of participants had to achieve a PFS2(Progression-Free Survival 2)/PFS1(Progression-Free Survival 1) ≥ 1.3 in a sample population of 25 evaluable patients. Sample size was calculated using an exact single-stage design for phase II studies with a one-sided type I error of 5% and a power of 90% under the assumption that PFS2/PFS1≥ 1.3 in ≤10% of patients would be clinically irrelevant, while a success rate ≥ 35% would merit further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or metastatic malignant solid tumors diagnosed by histology or cytology;
2. ECOG score 0-4 (3-4 points only for patients with tumor burden);
3. Those who fail or cannot tolerate standard treatment, or those who refuse standard treatment;
4. At least one measurable lesion that meets the RECIST 1.1 standard;
5. Expected survival period ≥ 3 months;
6. Age ≥ 18 years old;
7. Tumor tissue blocks with sufficient formalin fixed paraffin embedding (FFPE), or chest or ascites with cancer cells detected during treatment (not less than 200ml), or excised metastatic lymph nodes, or peripheral blood (approximately 5m1) can be used for genetic testing;
8. Understand and voluntarily participate in this study, and sign the informed consent form.

Exclusion Criteria:

1. Patients who have actively undergone or are currently participating in clinical trials for treatment;
2. Serious or uncontrolled medical diseases (i.e. uncontrolled diabetes, chronic kidney disease, chronic lung disease or uncontrolled active infection, mental diseases/social conditions that limit the compliance with the research requirements) that the researchers think will confuse the research treatment response analysis;
3. Pregnant or lactating patients, or any patients with fertility, have not taken appropriate pregnancy prevention measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
PFS2/PFS1(Progression Free Survival 2/Progression Free Survival 1) | 24 months
  The time to progression-free survival during the substudy (PFS2) exceeds the documented time to disease progression-free survival during the last treatment prior to substudy entry (PFS1) by at least 35% (ie, PFS2/PFS1≥1.3) or, if PFS1 is not evaluable, time to progressive disease exceeds 6 months.

SECONDARY OUTCOMES:
OS(Overall Survival) | 24 months
  Evaluation of overall survival (OS) defined as the time between inclusion and death, whatever the cause is. Alive patients will be censored at their last known contact date.
ORR(Objective Response Rate) | 24 months
  Evaluation of the best objective response rate (ORR) for each treatment according to RECIST 1.1. The best ORR is the best response reached during treatment according to RECIST 1.1 criteria.
Number of treatment related adverse events with grade 3 or greater severity by CTCAE 5.0 | 24 months
  Treatment related adverse events with grade 3 or greater severity by CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No